CLINICAL TRIAL: NCT04985929
Title: The Impact of the Vasodilator, Sildenafil, on the Pulmonary Circulation During Exercise in Healthy Trained and Untrained Humans
Brief Title: The Impact of Sildenafil on the Pulmonary Circulation in Healthy Trained and Untrained Humans
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: Pro000108975
Record Dates: First submitted 2021-07-23; First posted 2021-08-02 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Healthy
MeSH Terms: interventions — Sildenafil Citrate

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled cross-over design
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-blind, placebo-controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Healthy, Untrained (Experimental): Untrained participants will be defined as having a V̇O2peak of 30-45 ml.kg-1.min-1 and will be between 18-40 years of age.
  Interventions: Drug: Sildenafil 50 mg; Drug: Placebo
- Healthy, Trained (Experimental): Trained participants will be defined as having a V̇O2peak above 55 ml.kg-1.min-1 (females) and 60 ml.kg-1.min-1 (males) and will be between 18-40 years of age.
  Interventions: Drug: Sildenafil 50 mg; Drug: Placebo

INTERVENTIONS:
Drug: Sildenafil 50 mg — Sildenafil is a phosphodiesterase type-5 inhibitor, which augments/prolongs the naturally occurring nitric oxide mediated vasodilatory pathway. Sildenafil pill is over-encapsulated to be identical in appearance to the placebo intervention.
  Other Names: Accel-Sildenafil - 50 mg
Drug: Placebo — Medical-grade placebo pill, over-encapsulated to be identical in appearance to the sildenafil intervention.

SUMMARY:
There is emerging evidence suggesting that the pulmonary vasculature and right heart may play a role in the limitation of exercise capacity in healthy individuals. It is well established that aerobic training improves cardiovascular function. While the pulmonary system is integral to the function of the cardiopulmonary system, it has been traditionally accepted that lung function does not respond to exercise training. However, recent research suggests pulmonary vascular function adaptations may occur with aerobic training, and this may contribute to enhanced exercise tolerance. Research has highlighted that increased capillary blood volume (Vc) and diffusion capacity for carbon monoxide (DLCO) are correlated with higher cardiorespiratory fitness at rest. Additionally, endurance trained participants have increased exercise DLCO concomitant to higher resting Vc when compared to untrained participants, and during exercise this difference seems to be driven by higher membrane diffusing capacity (Dm), independent of Vc or VA (alveolar volume). Of importance is also the evidence that highlights endurance trained participants having reduced pulmonary arterial pressures at rest and during exercise. Reduced pulmonary arterial pressure in endurance trained participants despite endurance trained participants consistently displaying increased diffusion capacity/pulmonary perfusion at rest and during exercise suggests a lower threshold pressure for pulmonary capillary recruitment. Together, this cross-sectional evidence suggests improvements in the pulmonary circulation due to exercise training in order to facilitate gas exchange. Whether this apparent improvement in pulmonary circulation is due to enhanced pulmonary vascular function via NO mediated vasodilation must be determined experimentally. If sildenafil administration improves DLCO, Vc, and Dm, this would provide evidence that the NO mediated vasodilatory pathway plays a role in the regulation of vascular tone, function, and perfusion across the pulmonary vasculature. Should a larger response to sildenafil be observed in untrained persons, this would suggest better baseline vascular function in trained participants compared to untrained. This would provide strong evidence that aerobic training improves pulmonary vasculature function which is contrary to the conventional understanding of aerobic training on the cardiopulmonary system.

DETAILED DESCRIPTION:
Background

There is emerging evidence suggesting that the pulmonary vasculature and right heart may play a role in the limitation of exercise capacity in healthy individuals. It is well established that aerobic training improves cardiovascular function. While the pulmonary system is integral to the function of the cardiopulmonary system, it has been traditionally accepted that lung function does not respond to exercise training. However, recent research suggests pulmonary vascular function adaptations may occur with aerobic training, and this may contribute to enhanced exercise tolerance.

Research has highlighted that increased capillary blood volume (Vc) and diffusion capacity for carbon monoxide (DLCO) are correlated with higher cardiorespiratory fitness at rest. Additionally, endurance trained participants have increased exercise DLCO concomitant to higher resting Vc when compared to untrained participants, and during exercise this difference seems to be driven by higher membrane diffusing capacity (Dm), independent of Vc or VA (alveolar volume). Of importance is also the evidence that highlights endurance trained participants having reduced pulmonary arterial pressures at rest and during exercise. Reduced pulmonary arterial pressure in endurance trained participants despite endurance trained participants consistently displaying increased diffusion capacity/pulmonary perfusion at rest and during exercise suggests a lower threshold pressure for pulmonary capillary recruitment. Together, this cross-sectional evidence suggests improvements in the pulmonary circulation due to exercise training in order to facilitate gas exchange. Whether this apparent improvement in pulmonary circulation is due to enhanced pulmonary vascular function via NO mediated vasodilation must be determined experimentally. If sildenafil administration improves DLCO, Vc, and Dm, this would provide evidence that the NO mediated vasodilatory pathway plays a role in the regulation of vascular tone, function, and perfusion across the pulmonary vasculature. Should a larger response to sildenafil be observed in untrained persons, this would suggest better baseline vascular function in trained participants compared to untrained. This would provide strong evidence that aerobic training improves pulmonary vasculature function which is contrary to the conventional understanding of aerobic training on the cardiopulmonary system.

Some investigations on the pulmonary vasculature have been completed with the known pulmonary vasodilator, sildenafil. Sildenafil administration has been shown to reduce pulmonary artery pressure and improve exercise tolerance in normobaric hypoxic conditions in young healthy individuals. Further, one of these investigations determined sildenafil did not alter maximal oxygen consumption (V̇O2peak) in normoxia in moderately fit participants; however, this study was likely underpowered to detect a response. While some sildenafil interventional work has been conducted, no study to date has determined the effect of sildenafil on DLCO, Vc, and Dm during exercise in untrained vs. trained participants. If sildenafil administration improves DLCO, Vc, and Dm, this would provide evidence that the NO mediated vasodilatory pathway plays a role in the regulation of vascular tone, function, and perfusion across the pulmonary vasculature. Should a larger response to sildenafil be observed in untrained persons, this would suggest better baseline vascular function in trained participants compared to untrained. This would provide strong evidence that aerobic training improves pulmonary vasculature function which is contrary to the conventional understanding of aerobic training on the cardiopulmonary system.

Purpose

To examine the effects of the pulmonary vasodilator sildenafil on DLCO, Vc, and Dm in trained and untrained participants at rest and during exercise.

Hypothesis

If sildenafil administration improves DLCO, Vc, and Dm, this would provide evidence that the NO mediated vasodilatory pathway plays a role in the regulation of vascular tone, function, and perfusion across the pulmonary vasculature. Should a larger response to sildenafil be observed in untrained persons, this would suggest better baseline vascular function in trained participants compared to untrained. This would provide strong evidence that aerobic training improves pulmonary vasculature function which is contrary to the conventional understanding of aerobic training on the cardiopulmonary system.

Research Design

Randomized, double-blinded, placebo controlled cross-over design.

Trial Treatment

Treatment: Sildenafil (oral), 50 mg Placebo: Medical grade placebo pill

Duration

This randomized, double-blind, placebo controlled, cross-over, cross-sectional study will include 6 sessions and will be a crossover design with participants acting as their own controls. All exercise protocols will be conducted on an electronically braked cycle ergometer and will begin with a standardized warm-up and end with a standardized cool-down.

Session 1) During session 1, participants will provide informed consent and health screening (PAR-Q+), be familiarized to the laboratory and experimental measurement protocols, conduct a pulmonary function test, and conduct an incremental maximal exercise test to determine V̇O2peak on the cycle ergometer. A small blood sample will be collected via finger prick to measure hemoglobin (to correct DLCO). Specific relative workloads will be calculated cardiorespiratory and power output data obtained from the V̇O2peak protocol conducted during session 1.

Session 2 and 3) During sessions 2 and 3, participants will ingest either a placebo or 50 mg sildenafil, then rest a minimum of 30 minutes. Testing will start with measurement of resting diffusion capacity, pulmonary capillary blood volume (Vc), and membrane diffusion capacity (Dm) using the multiple fractional inspired oxygen (FIO2)-DLCO technique, with the order of FIO2 administration randomized and the participant in supine position. Supine DLCO measurements are to determine maximal resting DLCO and to quantify the impact of postural change on participant DLCO. Next, participants will complete resting baseline DLCO measurements seated on the cycle ergometer, followed by an absolute workload protocol with the exercise intensity set at 60 Watts for a duration of ten minutes. A small blood sample will be collected via finger prick to measure hemoglobin (to correct DLCO). During the absolute workload protocol, measurements will occur after the 4th minute of exercise, in order to allow verification of measurement equipment operation during exercise and to give the participant sufficient time to warm-up and hit steady state. Steady state will be defined as minute-by-minute change in heart rate ≤ 5 bpm. A minimum of 9 and no more than 12 breath-holds will be performed during this session. The order of sessions 2 and 3 will be randomized and the participant and laboratory technicians will be blinded to the administration of the pharmacological intervention.

Session 4 and 5) During sessions 4 and 5, participants will ingest either a placebo or 50 mg sildenafil, rest a minimum of 30 minutes, and then complete exercise DLCO sessions. The exercise DLCO sessions will include exercise intensities set at 30%, 60%, and 90% of individual V̇O2peak with the order of FIO2 administration and workload randomized. A minimum of 9 and no more than 12 breath-holds will be performed during this session. DLCO measurements will be taken after participants have attained steady-state at each workload. A small blood sample will be collected via finger prick to measure hemoglobin (to correct DLCO). Participants will complete active recovery (<100W) between workloads to minimize fatigue and metabolite accumulation similar to previous work. The order of sessions 4 and 5 will be randomized and the participant and laboratory technicians will be blinded to the administration of the pharmacological intervention.

Session 6) During session 6, participants will undergo echocardiography measurements at rest and during exercise after taking placebo and sildenafil. The order of drug administration during this session will not be randomized. Resting echocardiography will be conducted during quiet seated rest and exercise will be conducted exercising at 60 Watts, both on the same cycle ergometer.

Session 1 is anticipated to take ~2 hours. Sessions 2 and 3 are anticipated to take ~1.5 hours. Sessions 4 and 5 are anticipated to take 2 hours. Session 6 is anticipated to take 2 hours. The anticipated total study duration is ~11 hours. All sessions will be planned within a 6-week timeframe.

Statistical Methods

Data will be analyzed using commercially available software. A priori α = 0.05. Diffusion capacity response will be analyzed by group mean analysis with a two-way repeated measures ANOVA with the groupings as HI-FIT and LO-FIT (key variables DLCO, Dm, Vc) across all exercise intensities, consistent with previous work with similar methods and primary outcomes. Post-hoc testing will be conducted via Holm-Sidak method. The same approach will be used to determine differences in key variables from echocardiography (e.g. PASP).

ELIGIBILITY:
Inclusion Criteria:

* Untrained participants will be defined as having a V̇O2peak of 30-45 ml.kg-1.min-1.
* Trained participants will be defined as having a V̇O2peak above 55 ml.kg-1.min-1 (females) and 60 ml.kg-1.min-1 (males).
* All participants will be between the ages of 18-40 years.

Exclusion Criteria:

* Absolute contraindication to exercise testing or an orthopedic condition that may limit exercise testing as identified by standardized health screening tool (PAR-Q+).
* Pre-existing cardiac conditions (heart failure, congenital heart defect, valvular disease) that may limit exercise testing.
* A diagnosis of pulmonary hypertension.
* Current prescription drug use (excluding oral contraception for females).
* Pregnancy or lactation.
* Women of childbearing potential must be willing to use an acceptable method of contraception to avoid pregnancy throughout the study. Acceptable methods of contraception include tubal ligation, oral contraceptive, barrier methods (intra-uterine device, diaphragm, female condom, male condom). Abstinence is an acceptable form of contraception, only insofar as patients agree to use another acceptable method of birth control, preferably a barrier method, if they become sexually active.
* Postmenopausal female participants must be amenorrheic for ≥12 months.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2024-07-05 (Actual); Study Completion 2024-07-05 (Actual)

PRIMARY OUTCOMES:
Diffusion capacity of carbon monoxide (DLCO) | Minimum of 30 minutes post-dose.
  Diffusion capacity of carbon monoxide (DLCO) in selected body positions and exercise intensities. DLCO is measured with the Roughton-Forster Multiple FIO2 single-breath DLCO procedure.
Capillary blood volume (Vc) | Minimum of 30 minutes post-dose.
  Capillary blood volume is a component of DLCO and is measured with the Roughton-Forster Multiple FIO2 single-breath DLCO procedure.
Membrane diffusing capacity (Dm) | Minimum of 30 minutes post-dose.
  Membrane diffusing capacity is a component of DLCO and is measured with the Roughton-Forster Multiple FIO2 single-breath DLCO procedure.

SECONDARY OUTCOMES:
Pulmonary artery systolic pressure (PASP) | Minimum of 30 minutes post-dose.
  Pulmonary artery systolic pressure at rest and during exercise as determined via echocardiography.

CONTACTS AND LOCATIONS:
Overall Officials: Sean van Diepen, MD, Study Director — University of Alberta; Michael K Stickland, PhD, Principal Investigator — University of Alberta
Locations (1):
- Clinical Physiology Laboratory, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No
No IPD sharing plan.